CLINICAL TRIAL: NCT01834677
Title: Translational Research Evaluating Neurocognitive Memory Processes
Acronym: TREC-MP
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00039288; 5K23MH087739-03 (NIH)
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Neurocognition
Keywords: Depression; Neurocognition; Electroconvulsive Therapy (ECT); Parkinson's Disease
MeSH Terms: conditions — Depression; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy Human
- Depressed Human
- Depressed Human, Undergoing Electroconvulsive Therapy: Electroconvulsive Therapy is being received as standard of care, not as a study intervention.
- Human Diagnosed with Parkinson's Disease

SUMMARY:
The purpose of this study is to evaluate the psychometric properties and utility of new, computerized, neurocognitive measures in humans with depression, and humans with depression undergoing electroconvulsive therapy (ECT). The benefits of the study outweigh the risk as there is the possibility of developing better computerized neurocognitive measures, and the risks are limited to no more than minimal test related fatigue and psychological stress.

Depressed humans, depressed human participants undergoing ECT, and humans diagnosed with Parkinson's disease (age 18-85) will be invited to participate in this study. After providing informed consent participants will undergo a clinical psychiatric evaluation to confirm the inclusion/exclusion criteria. After the clinical psychiatric evaluation, participants will complete common and new neurocognitive measures. There will be a total of two testing visits (baseline, 1-month follow-up). The anticipated duration of the participant's involvement is no more than 2 study visits that can take place over a 4-day period (i.e., the clinical evaluation can occur on day 1 and the neuropsychological measures can be administered on day 2 of each study visit) equating to approximately 6-hours (3-hours each day) per study visit.

ELIGIBILITY:
Inclusion Criteria:Depressed Individuals

1. Male and female subjects, age 18-85
2. DSM-IV-TR diagnosis of major depressive episode, unipolar, confirmed by the MINI-PLUS [221]
3. HRSD24 total score > 10
4. MMSE total score > 26
5. Graduated from high school
6. Competent to provide informed consent

Inclusion Criteria:Depressed Individuals Receiving ECT

1. Same as for Depressed Cohort Inclusion Criteria (see above)
2. Referred for ECT
3. Subject competent to provide informed consent

Inclusion Criteria:Individuals Diagnosed with PD

1. Male and female subjects, age 18-85
2. Diagnosed with PD
3. MMSE total score > 20
4. Graduate high school
5. Subject competent to provide informed consent

Exclusion Criteria:Depressed Individuals/Depressed Individuals Receiving ECT

1. Lifetime history of bipolar disorder, schizophrenia, schizoaffective disorder, or mental retardation
2. Current neurostimulation treatment (e.g., ECT, MST, rTMS, vagus nerve stimulation, deep brain stimulation)
3. Current alcohol abuse or dependence within past 12 months
4. Current substance abuse or dependence within past 12 months
5. Lifetime mental retardation
6. History of central nervous system (CNS) disease
7. Current diagnosis of dementia or delirium
8. Current visual, auditory, or motor impairment that compromises ability to take tests
9. Unable to read or comprehend English

Exclusion Criteria:Individuals Diagnosed with PD

1. Lifetime history of bipolar disorder, schizophrenia, schizoaffective disorder, or mental retardation
2. Current neurostimulation treatment (e.g., ECT, MST, rTMS, vagus nerve stimulation, deep brain stimulation)
3. Current alcohol abuse or dependence within past 12 months
4. Current substance abuse or dependence within past 12 months
5. Lifetime mental retardation
6. History of central nervous system (CNS) disease other than Parkinson's Disease
7. Current diagnosis of dementia or delirium
8. Current visual, auditory, or motor impairment that compromises ability to take tests
9. Unable to read or comprehend English

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are able to contact the study team. The depressed ECT cohort will be referred to study team.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2013-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
California Verbal Learning Test-II | Baseline
  The California Verbal Learning Test-II (CVLT-II) is a standard neuropsychological instrument that assesses verbal learning and memory.
California Verbal Learning Test-II | 1-Month Follow-up
  The California Verbal Learning Test-II (CVLT-II) is a standard neuropsychological instrument that assesses verbal learning and memory.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn McClintock, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Universtiy Medical Center, Durham, North Carolina, United States